CLINICAL TRIAL: NCT03585855
Title: Autologous Mesenchymal Stem Cell Transplantation in the Treatment of Chronic Antibody Mediated Kidney Graft Rejection (ABMR)
Brief Title: Mesenchymal Stem Cell Transplantation in the Treatment of Chronic Antibody Mediated Kidney Graft Rejection (ABMR)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety reasons
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Veceric-Haler Zeljka, Principal investigator, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P3-0323
Record Dates: First submitted 2018-06-25; First posted 2018-07-13 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Interventional

STUDY DESIGN:
Intervention Model Description: comparison with historic control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historic control (No Intervention): historic cohort of patients with ABMR treated with standard of care therapy
- MSC transplantation (Experimental): patients with ABMR treated with MSC transplantation
  Interventions: Other: MSC transplantation

INTERVENTIONS:
Other: MSC transplantation — MSC transplantation: patients with ABMR treated with MSC transplantation
  Arms: MSC transplantation

SUMMARY:
Transplant rejection is one of the biggest limitations in renal transplant procedures, where the kidney can undergo an acute, late acute, or chronic transplant rejection. With the advancement in transplantation protocols, acute survival of renal transplants has improved, but long-term survival is still unsatisfactory, as most of the renal transplants develop chronic graft rejection. Unfortunately, there is little the investigators know when it comes to improving long-term survival of renal transplants. Mesenchymal stem cells (MSC) have been shown to have immunosuppressive and repairing properties. The purpose of this study is to find out whether MSC in combination with standard therapy of antibody mediated rejection (ABMR) are more effective in preventing organ deterioration and maintaining kidney function.

DETAILED DESCRIPTION:
Participants will be assigned to receive the full immunosuppressive therapy indicated to treat chronic ABMR (including plasmapheresis (PF) 7x, intravenous immune globulins 100 mg/kg 7x, corticosteroid) and MSC infusions (2x106cells/kg bw after PF) (Group 1) and be compared to historic controls according to "propensity score matching" (treated with immunosuppressive therapy alone (Group 2)). Patients will undergo MSC infusions at the start of the study after each PF. One year post- infusions, patients will be evaluated and undergo kidney biopsies. Blood collection will occur at regular intervals, serum creatinine and the estimated creatinine clearance will be monthly recorded. The transplanted kidney function and morphology (US Doppler) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a renal allograft, male and female patients age >18
* The eGF>20 ml/min/1.73 m2,
* Renal biopsy Criteria: chronic active ABMR.
* Written informed consent, compliant with local regulations.

Exclusion Criteria:

* Recipients of multiple organs.
* Pregnant women.
* Malignant disease in last 5 years
* Active autoimmune disease
* Active infection including hepatitis B, hepatitis C, HIV, or tuberculosis
* Evidence of congestive cardiac failure and/or acute coronary syndrome in past 6 months.
* Evidence of liver disease
* Inadequate compliance to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Safety of MSC transplantation as assessed by adverse events according to CTCAE Version 5Estimated glomerular filtration rate (eGFR) | 12 months
  Adverse events according to CTCAE Version 5

SECONDARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | 12 months
  eGFR at up to 12 months post MSC transplantation
Graft survival rate | 12 months
  Graft survival rate at 12 months post MSC transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Željka Večerić-Haler, MDPhD, Principal Investigator — assist.prof.Željka Večerić-Haler, MDPhD
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
12 months